CLINICAL TRIAL: NCT06653517
Title: Neoadjuvant BRAFV600E-Targeted Therapy for Conventional Ameloblastoma of the Jaw:A Single-Arm Clinical Study
Brief Title: Clinical Study of Neoadjuvant Targeted Therapy for Ameloblastoma
Acronym: NETCAM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NETCAM_2024CT
Record Dates: First submitted 2024-10-15; First posted 2024-10-22 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Ameloblastoma; BRAF V600E Mutation Positive
Keywords: Dabrafenib; Trametinib; BRAF V600E Mutation; Conventional Ameloblastoma; Preoperative Targeted Induction Therapy; Mandibular Continuity-Preserving Surgery; Non-radical Resectable Surgery
MeSH Terms: conditions — Ameloblastoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dabrafenib and Trametinib Treatment Arm (Experimental): Dabrafenib: 150 mg twice daily, not to be taken if less than 6 hours remain to the next dose.
  Trametinib: 2 mg once daily, not to be taken if less than 12 hours remain to the next dose.
  Cycle Length: 30 days. Initial Follow-Up: After each of the first two cycles. Toxicity Management: Discontinue if intolerable toxicity occurs. Long-Term Follow-Up: Every two cycles. Criteria for Surgery: Confirmed by at least two chief physicians.
  Interventions: Drug: Dabrafenib; Drug: Trametinib

INTERVENTIONS:
Drug: Dabrafenib — Dosage: 150 mg orally, twice daily (total daily dose of 300 mg) Administration: Administer at approximately 12 hours apart. Take at the same time each day. If a dose is missed and less than 6 hours remain until the next dose, skip the missed dose. Do not open, crush, or break the capsules.
  Usage in Combination: When used in combination with trametinib, trametinib should be taken once daily at the same time as either the morning or evening dose of dabrafenib to ensure synchronization of the treatment schedule.
  Other Names: Tafinlar
Drug: Trametinib — Dosage: 2 mg orally, once daily Administration: Administer at least 1 hour before or 2 hours after a meal. Take at the same time each day. If a dose is missed, it should be taken no later than 12 hours before the next scheduled dose; otherwise, skip the missed dose.
  Usage in Combination: When used in combination with trametinib, trametinib should be taken once daily at the same time as either the morning or evening dose of dabrafenib to ensure synchronization of the treatment schedule.
  Other Names: Mekinist

SUMMARY:
This study aims to evaluate the tumor shrinkage effect of preoperative targeted induction therapy with dabrafenib and trametinib in patients with conventional ameloblastoma harboring the BRAF V600E mutation. The study will assess the proportion of cases where mandibular continuity cannot be preserved that can be converted to cases where mandibular continuity is preserved, as well as the proportion of cases where complete resection is initially not feasible that become resectable.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Ⅰ. To observe the proportion of patients with ameloblastoma requiring mandibular segmental resection at initial diagnosis who can convert to mandibular preservation surgery after preoperative induction therapy with dabrafenib and trametinib.

Ⅱ.To observe the proportion of cases initially deemed non-radical resectable Surgery that become resectable

SECONDARY OBJECTIVES:

Ⅰ. Radiological response Ⅱ. Pathological response Ⅲ. Local recurrence-free survival(LRFS) Ⅳ.Feasibility and safety in this patient population

OUTLINE:

Dabrafenib:

Dosage: 150 mg twice daily (total daily dose of 300 mg). Administration: Must be taken in combination with trametinib until disease progression or intolerable toxicity occurs. Administer at least 1 hour before or 2 hours after a meal, with approximately 12 hours between doses. Take at the same time each day. If a dose is missed and less than 6 hours remain until the next dose, the missed dose should not be taken. When used in combination with trametinib, take trametinib once daily at the same time as the morning or evening dose of dabrafenib. Do not open, crush, or break the capsules.

Trametinib:

Dosage: 2 mg once daily orally, in combination with dabrafenib, until disease progression or intolerable toxicity occurs.

Administration: Administer at least 1 hour before or 2 hours after a meal. Take at the same time each day. If a dose is missed, it should be taken no later than 12 hours before the next scheduled dose. If less than 12 hours remain until the next dose, the missed dose should not be taken. When used in combination with dabrafenib, take trametinib once daily at the same time as the morning or evening dose of dabrafenib. Do not chew or crush the tablets.

Treatment Cycle:

Cycle Length: Each cycle lasts 30 days. Initial Follow-Up: Follow-up after each of the first two cycles with a consultation, physical examination, imaging studies, and relevant laboratory tests to evaluate drug toxicity, safety, and tumor shrinkage rate.

Adjustment and Transition to Surgery:

Toxicity Management: If intolerable drug toxicity or adverse reactions occur that cannot be managed by dose adjustment, discontinue treatment immediately and switch to traditional surgical treatment.

Post Two-Cycles Evaluation: After the first two cycles, if intolerable adverse reactions persist or the tumor continues to progress despite dose adjustments, switch to traditional surgical treatment. If the tumor does not progress, continue long-term medication.

Long-Term Treatment Follow-Up:

Follow-Up Schedule: Conduct follow-up evaluations every two cycles, including consultations, physical examinations, imaging studies, and relevant laboratory tests to evaluate drug toxicity, safety, and tumor shrinkage rate.

Criteria for Surgery: If tumor shrinkage reaches a plateau or the patient meets the criteria for mandibular preservation surgery, and the surgical plan is confirmed independently by at least two chief physicians in the department, record this in the case report form and discontinue the medication in preparation for scheduled surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years;
2. Diagnosed with solid/multicystic type ameloblastoma with confirmed BRAF V600E mutation by next-generation sequencing (NGS);
3. Requires mandibular segmental resection at diagnosis, confirmed by two or more chief physicians;
4. No distant metastasis or malignancy;
5. ECOG score 0-1;
6. Willing to undergo surgery after induction therapy;
7. No significant contraindications to MEK and BRAF inhibitors;
8. Major organ function meets the following standards:

   1. Hematological: WBC ≥ 4.0×10^9/L, ANC ≥ 1.5×10^9/L, PLT ≥ 100×10^9/L, Hb ≥ 90g/L (no transfusion or blood products, no use of G-CSF or other hematopoietic stimulants within 14 days);
   2. Biochemical: Serum albumin ≥ 3.0 g/dL, TBIL ≤ 1.5×ULN, ALT/AST ≤ 2.5×ULN, BUN/CRE ≤ 1.5×ULN or creatinine clearance rate ≥ 60 ml/min;
   3. Coagulation: INR or PT ≤ 1.5×ULN (anticoagulant-treated subjects must have PT within the intended range);
9. Women of childbearing age must use effective contraception, have a negative pregnancy test within 7 days before enrollment, and agree to use effective contraception during the study and for 16 weeks after the last dose of trametinib and dabrafenib. Male subjects with partners of childbearing age must use effective contraception during the study and for 16 weeks after the last dose of trametinib and dabrafenib.
10. Voluntary participation with signed informed consent, good compliance, and cooperation for follow-up.

Exclusion Criteria:

1. Previous use of dabrafenib, trametinib, or other BRAF/MEK inhibitors;
2. Active autoimmune diseases (stable conditions not requiring systemic immunosuppression allowed);
3. Congenital or acquired immunodeficiency (e.g., HIV), active hepatitis B (HBV-DNA ≥ 10^4 copies/ml), or hepatitis C (positive HCV antibody and HCR-RNA above the detection limit);
4. Known allergy to study drugs or their excipients, or severe allergic reactions to other monoclonal antibodies or targeted drugs;
5. Myocardial infarction, severe/unstable angina, NYHA class II or higher heart failure, significant arrhythmias, or symptomatic congestive heart failure within 6 months before enrollment;
6. Live vaccination within 4 weeks before the first dose of study drugs (inactivated virus vaccines allowed for seasonal flu, but live attenuated intranasal vaccines not allowed);
7. History of allogeneic organ or hematopoietic stem cell transplantation;
8. Known history of substance abuse or drug addiction;
9. Pregnant or breastfeeding women;
10. Diagnosed with any other tumors within 5 years before the study, except for locally treatable and cured basal cell carcinoma, squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, ductal carcinoma in situ, papillary thyroid carcinoma, and benign tumors;
11. Other severe physical or mental diseases or laboratory abnormalities that may increase the risk of participation or interfere with study results, deemed unsuitable for participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Eligible for Mandibular Continuity-Preserving Surgery | After completion of two 30-day cycles of therapy (approximately 2 months)
  The proportion of patients initially requiring mandibular segmental resection who become eligible for mandibular continuity-preserving surgery after preoperative targeted induction therapy with dabrafenib and trametinib.
Proportion of Non-radical Resectable Cases Becoming Resectable | After completion of two 30-day cycles of therapy (approximately 2 months)
  The proportion of patients initially deemed non-radical resectable who become resectable after completing two cycles of preoperative targeted induction therapy with dabrafenib and trametinib.

SECONDARY OUTCOMES:
Radiological Response | After completion of two 30-day cycles of therapy (approximately 2 months)
  The evaluation of tumor response using radiological studies such as MRI or CT scans after preoperative targeted induction therapy with dabrafenib and trametinib.
Pathological Response | After completion of two 30-day cycles of therapy (approximately 2 months)
  The assessment of tumor pathological changes after preoperative targeted induction therapy with dabrafenib and trametinib, based on biopsy or surgical specimens.
Local Recurrence-Free Survival (LRFS) | 3 months
  The time from the start of treatment to the occurrence of local recurrence or death from any cause, whichever occurs first.
Adverse Effects and Safety | Throughout the study period, up to 12 months
  The incidence and severity of adverse effects related to the combination therapy with dabrafenib and trametinib, assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: CAO Wei, PHD;MD, Principal Investigator — Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China